CLINICAL TRIAL: NCT02571374
Title: Change in Incidence of Surgical Site Infection After Resection of Colorectal Cancer Between Patients Receiving a Symbiotic Compound and Patients Receiving a Placebo.
Brief Title: Symbiotics to Prevent Postoperative Infection in Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline Gamarra Taborda, ms, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: symbioticcolorectalcancer
Record Dates: First submitted 2014-04-11; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer; Surgical Site Infection
Keywords: symbiotic; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- symbiotic group (Experimental): Symbiotic group
  Interventions: Dietary Supplement: symbiotic group
- placebo group (Placebo Comparator): placebo group
  Interventions: Dietary Supplement: placebo group

INTERVENTIONS:
Dietary Supplement: symbiotic group — this group received sachets of symbiotic
  Arms: symbiotic group
Dietary Supplement: placebo group — this group received placebo
  Other Names: maltodextrina
  Arms: placebo group

SUMMARY:
This is a double blind randomized trial in which patients with colorectal cancer undergoing surgery will be selected to receive either a symbiotic formulation or placebo. The researchers will compare incidence of surgical site infection between the study groups.

DETAILED DESCRIPTION:
This is a double blind randomized trial in which patients with colorectal cancer undergoing surgery will be randomly selected to receive either a symbiotic formulation or placebo during the perioperative period. The researchers will compare incidence of surgical site infection, detected by clinical examination and complementary tests (CT scans, X-rays, microbiological and hematological tests) between the study groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 85 years old;
* Colorectal cancer patients.
* Ability to understand and signing the informed consent

Exclusion Criteria:

* Pregnancy (early diagnosis)
* Reduced intellectual level that could prevent proper understanding of the objectives of the study
* Patients with rectal cancer undergoing neoadjuvant treatment (chemotherapy and radiotherapy)
* Use of products with prebiotic, probiotic and / or symbiotic function or fiber module; by more than 3x a week
* Refusal to participate and / or to sign the Consent Form Free and Clear

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with colorectal cancer on symbiotic to prevent postoperative infection | 1 month
  This is a double blind randomized trial in which patients with colorectal cancer undergoing surgery will be selected to receive either a symbiotic formulation or placebo. After we will compare the number of participants with incidence of surgical site infection between the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Taborda, ms, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil